CLINICAL TRIAL: NCT06777433
Title: An Open-Label, Single Dose, Single Arm, Multicenter Phase 2b Study to Establish the Imaging Performance of RAD101 Positron Emission Tomography (PET) in Participants With Suspected Recurrent Brain Metastases From Solid Tumors
Brief Title: Phase 2b Imaging Study of RAD101 in Participants With Suspected Recurrent Brain Metastases
Acronym: RAD101
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Radiopharm Theranostics, Ltd (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCP-PRT-101-001
Record Dates: First submitted 2024-12-19; First posted 2025-01-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-03

CONDITIONS: Brain Metastases From Solid Tumors
Keywords: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAD101 (18F-Fluorescence polarization immunoassay (FPIA)) (Experimental): 370 MBq (10 mCi) single dose administered at Day 1 visit
  Interventions: Drug: RAD101 (18F-FPIA)

INTERVENTIONS:
Drug: RAD101 (18F-FPIA) — A single dose of 18F-RAD101 with a maximum of 370 MBq (10 mCi) administered as a slow IV bolus injection over a maximum of 30 seconds, followed by a saline flush.

SUMMARY:
This is an open-label, single dose, single arm, multicenter Phase 2b study to establish the imaging performance of RAD101 PET in participants who are ≥ 18 years of age and with suspected recurrent brain metastases from solid tumors.

The study consists of a 4-week Screening Period, a 3-day Imaging and Safety Follow-Up Period, and a Data Collection Period of up to 6 months. Participant eligibility will be determined during the Screening Period and eligible participants will be enrolled in the study. On Day 1, the enrolled participants will receive a single dose of the investigational medicinal product (IMP), RAD101. Participants will then proceed with a whole brain PET scan. A high-resolution Magnetic Resonance Imaging (MRI) will be performed in joint acquisition with PET or separately on the same day, or on the day prior to or the day following RAD101 administration. For applicable study sites where PK samples will be collected, whole body PET scans will be performed, blood samples will be drawn, and urine will be collected throughout the scanning period. A phone follow-up will be performed on Day 3 (+ 1 day). Participants will have follow-up (longitudinal) MRI (otherwise CT) scans (longitudinal imaging) and/ or a biopsy according to their Standard of Care (SoC). The longitudinal image results, and details of the biopsy if performed as part of SoC (i.e., location and histopathology results), will be collected during the 6- month Data Collection Period.

DETAILED DESCRIPTION:
This is an open-label, single dose, single arm, multicenter Phase 2b study to establish the imaging performance of RAD101 PET in participants who are ≥ 18 years of age and with suspected recurrent brain metastases from solid tumors. Approximately 30 participants will be enrolled in the study. To avoid overrepresentation of a specific tumor type, a maximum of 15 participants per tumor type will be enrolled: lung, breast, colon, kidney, or melanoma.

The study consists of a 4-week Screening Period, a 3-day Imaging and Safety Follow-Up Period, and a Data Collection Period of up to 6 months. Participant eligibility will be determined during the Screening Period and eligible participants will be enrolled in the study. All participants will have a post-SRS (stereotactic radiosurgery)/ SRT (stereotactic radiotherapy) MRI (otherwise CT) performed as their SoC within 8 weeks before Day 1. For enrolled participants, the screening MRI (otherwise CT) images will be collected and submitted for central imaging review. On Day 1, the enrolled participants will receive a single dose of the investigational medicinal product (IMP), RAD101, at a target dose of 370 Megabecquerel (MBq) (10 millicurie (mCi)) ± 10% through a slow intravenous (IV) bolus injection over a maximum of 30 seconds, followed by a saline flush. Participants will then proceed with a whole brain PET scan at 60 ± 10 min post-dose. A high-resolution MRI will be performed in joint acquisition with PET or separately on the same day, or on the day prior or the day following RAD101 administration. For applicable study sites where PK samples will be collected, whole body PET scans will be performed, blood samples will be drawn, and urine will be collected throughout the scanning period. Safety assessments, such as physical examination, vital signs, Electrocardiogram (ECG), and laboratory tests, will be conducted on Day 1 before RAD101 administration. Vital signs and ECG will be repeated at the end of infusion (for participants undergoing PK assessments) 35 ± 5 min following RAD101 administration on Day 1. A phone follow-up will be performed on Day 3 (+ 1 day).

Participants will have follow-up (longitudinal) MRI (otherwise CT) scans (longitudinal imaging) and/ or a biopsy according to their SoC. If a biopsy is performed as part of their SoC during follow-up, the location of the biopsied lesion(s) and results of histopathology assessments on the lesion(s) will be collected. The longitudinal image results will be collected for central reading until a SoC biopsy is performed and the histopathology results are available, or up to 6 months following RAD101 administration, whichever comes first. The longitudinal image results, and details of the biopsy if performed as part of SoC (i.e., location and histopathology results), will be collected during the 6- month Data Collection Period.

To limit the number of participants being exposed to a dose-ranging study, the minimum effective dose (MBq) of RAD101 will be assessed on a subset of 6 to 10 participants using images obtained by simulated count reduction.

The duration of study participation for each participant is approximately 211 days (7 months), including 28 days of the Screening Period, 3 days of the Imaging and Safety Follow-Up Period, and up to 180 days of the Data Collection Period. The duration of the entire study is planned to be approximately 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 18 years of age at the time of signing the informed consent.
2. Participant has one of the following histopathologically confirmed advanced solid tumors with known history of brain metastases: lung, breast, colon, kidney, or melanoma, and with known history of brain metastases. Other primary tumor diagnoses may be approved on a case-by-case basis following discussion with the Sponsor.
3. Participant has undergone SRS or SRT for their brain metastases prior to study screening with pre-planning images available for submission to the centralized imaging reader as reference.
4. Participant has suspected but not confirmed recurrent brain metastases in at least 1 lesion previously treated with SRS or SRT, based on gadolinium-enhanced volumetric MRI (MRI preferred, otherwise CT) within 8 weeks prior to Day 1, with post-SRS/SRT images available for submission to the centralized imaging reader as reference. If the SoC scan was performed > 8 weeks before Day 1, discussion with the Sponsor is required to determine eligibility. In addition, each suspected lesion must meet the following criteria:

   1. Size must be at least 5 mm in longest diameter seen on 2 slices on the volumetric MRI analyzed at 2.5 mm slice thickness, AND
   2. Lesion does not meet complete response criteria or unequivocal progressive disease criteria in the medical opinion of the evaluating provider or as outlined in Appendix 5 (Section 10.5).

   Note: New brain metastases or new leptomeningeal disease based on macrocyclic gadolinium-enhanced MRI within 6 weeks prior to Day 1, in addition to the above findings, are permitted.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
6. Estimated glomerular filtration rate (eGFR) calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula and individualized for participant's body surface area (BSA) ≥ 45 ml/min (ie, nonindexed GFR = indexed GFR × BSA (m2)/1.73 m2)
7. Life expectancy ≥4 months
8. Participant is not scheduled to undergo a confirmatory biopsy to characterize MRI findings until after the Day 1 study procedures have been completed.
9. Female participants must meet either of the following criteria:

   1. Women of childbearing potential (WOCBP) must have a negative beta human chorionic gonadotropin (β-hCG) test within 72 hours before administration of IMP and must not be breastfeeding. WOCBP, defined as all women physiologically capable of becoming pregnant, should agree to use highly effective methods of contraception during dosing and for 12 hours after administration of RAD101.
   2. Women who are not of childbearing potential are those who are surgically sterile or post-menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
10. Male participants who are able to father a child must agree to avoid impregnating a partner and to adhere to a highly effective method of contraception during dosing and for 12 hours after administration of IMP. All male participants must agree to not donate sperm for 12 hours after administration of IMP.

    Highly effective contraception methods include:
    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (i.e., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Female sterilization (have had bilateral surgical oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
    3. Male sterilization (at least 6 months prior to Screening). The vasectomized male partner should be the sole partner for that participant and the absence of sperm should be confirmed.
    4. Use of oral, injected, or implanted hormonal methods of contraception, or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that inhibit ovulation and have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking IMP. Acceptable contraception methods are further described in the protocol.
11. Willing and capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF), and willing to comply with all study procedures.

Exclusion Criteria:

1. History of known additional malignancy that is progressing or requires treatment.
2. Brain surgery for the target lesion within 4 weeks before the screening MRI.
3. Whole brain Radiation Therapy (RT), SRT, or SRS within 6 weeks of Day 1
4. Baseline Fridericia-corrected QT interval (QTcF) > 470 msec or history of congenital long QT syndrome
5. Any medical condition that would, in the Investigator's judgment, prevent the participant's full participation in the clinical study due to safety concerns or compliance with clinical study procedures, such as participants with severe claustrophobia who are unresponsive to oral anxiolytics, participants with low back pain who cannot lie comfortably on an imaging table, and participants who are hyperactive or hyperkinetic such that they cannot tolerate lying still for multiple time point imaging procedures.
6. Participation in any other investigational trial from the time of informed consent signature to the end of the Imaging and Safety Follow-Up Period if participation in the other study would interfere with the current study or would not be allowed by the other study. Participation in another study should be discussed with the Sponsor.
7. History of uncontrolled allergic reactions and/or known or expected hypersensitivity to RAD101, or any of its excipients, and/or macrocyclic gadolinium-based contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Concordance between RAD101 PET/MRI and MRI with macrocyclic gadolinium | 1 Week
  Number, size, and proportion of SRS/SRT-treated lesions identified by both RAD101 PET/MRI and MRI (with macrocyclic gadolinium)
Concordance between RAD101 PET/MRI and MRI with macrocyclic gadolinium | 1 Week
  Number, size, and proportion of SRS/SRT-treated lesions identified by RAD101 PET/MRI and not identified by MRI (with macrocyclic gadolinium)
Concordance between RAD101 PET/MRI and MRI with macrocyclic gadolinium | 1 Week
  Number, size, and proportion of SRS/SRT-treated lesions not identified by RAD101 PET/MRI and identified by MRI (with macrocyclic gadolinium)

SECONDARY OUTCOMES:
Accuracy of RAD101 in identifying tumor recurrence versus radiation necrosis in previously SRS-treated brain metastasis | 6 months
  Standard of care imaging using longitudinal MRI scans or histopathology based on RANO-BM response criteria
Safety and tolerability of a single dose of RAD101 | 48 Hours
  The properties, incidence, nature and severity of AEs and SAEs per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Optimal dose of RAD101 | 1 week
  Activity (MBq) of RAD101 in images obtained by simulated count reduction
Performance of RAD101 PET in identifying tumor lesions | 1 week
  Maximum standardized uptake values (Standardized uptake value (SUV)max) in suspected tumor lesions
Performance of RAD101 PET in identifying tumor lesions | 1 week
  Mean standardized uptake value (SUVmean) in tumor lesions
Performance of RAD101 PET in identifying tumor lesions | 1 week
  Lesion SUVmean to normal brain SUVmean ratio
Performance of RAD101 PET in identifying tumor lesions | 1 week
  Lesion SUVmax to normal brain SUVmax ratio

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Voliotis, MD, Study Director — Radiopharm Theranostics
Locations (5):
- United States (5):
  - Ascension Illinois Oncology Research, Hoffman Estates, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - BAMF Health, Grand Rapids, Michigan

IPD SHARING:
Plan to Share IPD: No